CLINICAL TRIAL: NCT01358487
Title: Internet Intervention to Prevent Major Depressive Episodes
Brief Title: Healthy Mood Internet Intervention Research Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHR10-00059; 1R34MH091231-01 (NIH)
Record Dates: First submitted 2010-10-12; First posted 2011-05-23 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Major Depression
Keywords: Major depression; Cognitive Behavioral preventive intervention; Mood Management; Self-help; Internet
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online self-help mood management course (Active Comparator): Online self-help mood management course based on cognitive behavioral therapy and social cognitive theory, plus automated online follow ups using email reminders and incentives for completing follow-ups
  Interventions: Behavioral: Online + incentives Follow-up Group
- Online self-help course plus live follow-up if needed (Experimental): Intervention and automated follow ups with incentives as in the active comparator condition. The experimental procedure is adding live phone follow-ups if participant does not complete online assessment surveys at 1, 3, and 6 months in response to automated emails.
  Interventions: Behavioral: Online self-help course plus live follow-up if needed

INTERVENTIONS:
Behavioral: Online self-help course plus live follow-up if needed — In addition to the self-help mood management course and the email reminders to return to the site to complete assessments at 1, 3, and 6 months (and the monetary incentives), this condition will also receive phone reminders if they do not complete assessments online.
  Arms: Online self-help course plus live follow-up if needed
Behavioral: Online + incentives Follow-up Group — This group tests online email reminders and monetary online incentives to estimate percentage of participants who will complete online assessments at 1, 3, and 6 month follow-ups.
  Arms: Online self-help mood management course

SUMMARY:
The purpose of the study is:

1. to study whether individuals WHO ARE NOT CURRENTLY SERIOUSLY DEPRESSED will participate in an online study to prevent clinical depression and
2. to estimate the percentage of participants who will complete online assessments at 1, 3, and 6 months when receiving either a) email reminders + monetary online incentives or b) email reminders + monetary incentives + phone calls.

NOTE: RECRUITMENT IS COMPLETED.

DETAILED DESCRIPTION:
In 2002, NIMH released an initiative that called upon researchers to improve psychosocial interventions for unipolar and bipolar depression. The Workgroup charged with this task recommended that researchers consider the "development of interventions that PREVENT onset and recurrence of clinical episodes in at-risk populations and [the] development of user-friendly interventions and nontraditional delivery methods to increase access to evidence-based interventions" (Hollon et al., 2002, p. 610). The overall goal of this research program aims to address these two priorities by adapting an empirically-validated depression intervention to the Internet. The current research study will eventually provide an online site to study whether clinical episodes of depression can be prevented by making the online Website available to people who are NOT currently depressed, but may be at risk for depression.

Study 1: the NIMH-funded pilot study. For Study 1, the investigators will conduct usability testing with 60 participants (half English-speaking and half Spanish-speaking) recruited at San Francisco General Hospital with the sole purpose of providing feedback on the Healthy Mood Management Project Website being developed. The investigators will not be testing the intervention itself on these usability testing participants.

The investigators will then recruit 150 participants (half English-speaking [NOW COMPLETED] and half Spanish-speaking [STILL RECRUITING]) WHO ARE NOT CURRENTLY DEPRESSED to use the Healthy Mood Management Project Website online. In this part of the study the investigators will compare follow-up completion rates obtained by (email reminders + monetary incentives) versus (email reminders + monetary incentives + phone call follow-ups). All participants will get automatic email reminders with links to return to the study site to fill out FU surveys at 1, 3, and 6 months. All participants will also be offered monetary incentives that can be obtained online. In addition, half of the participants (chosen at random) will receive phone calls if they do not complete follow-up surveys online. This will allow us to determine whether the phone call follow-ups significantly improve follow-up rates.

The monetary incentives will be provided as online gift certificates to Amazon.com. The incentives will be provided by sending the participant a code which allows the user to purchase products (books, etc.) up to the amount provided.

The two groups to be compared are:

1. Email reminders + incentives
2. Email reminders + incentives + phone calls (to collect data if not done online)

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* regular (>1 time/week) access to internet and email,
* valid email address
* fluent or almost fluent in English or Spanish [NOTE: ENGLISH RECRUITMENT COMPLETED. SPANISH RECRUITMENT CONTINUES]
* looking for information to help themselves, rather than another person
* must complete screening survey at the following Website: https://ihrc.ucsf.edu/Collector/Survey.ashx?Name=DPC_ScreenSurvey&SOURCE=Prev4

Exclusion Criteria:

* less than 18 years of age
* sporadic (<1 time/week) access to internet and email
* no valid email address
* not fluent in English or Spanish
* looking for information to help someone else
* currently suffering from serious depression and/or in treatment for depression (If you are currently depressed, consider applying for a related Internet study to manage serious depression symptoms by going to the following Website: https://ihrc.ucsf.edu/interventionConsole/Default.aspx?ConsoleName=DepressionManagementCourse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
PHQ-9 | Baseline, 1, 3, and 6 months post consent
  Screens for symptoms of major depressive episodes (MDE).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F. Muñoz, Ph.D., Principal Investigator — UCSF/SFGH
Locations (1):
- University of California, San Francisco, San Francisco, California, United States